CLINICAL TRIAL: NCT07173660
Title: Consensus Statements on Deep Brain Stimulation in Patients With Parkinson's Disease - A Delphi Study
Brief Title: Consensus Statements on Deep Brain Stimulation in Patients With Parkinson's Disease
Acronym: DBS_Consensus
Status: Not yet recruiting | Type: Observational
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Prof. Dr, University Magna Graecia
Other Study IDs: DBS Consensus
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Deep Brain Stimulation; Parkinson Disease
Keywords: Expert Consensus; Neurosurgery
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expert Panel: An Italian expert panel of about 30 healthcare professionals, including neurosurgeons with expertise in deep brain stimulation for patients with Parkinson's disease.
  Interventions: Other: Delphi study

INTERVENTIONS:
Other: Delphi study — A Delphi study will be conducted with several rounds up to stable expert consensus or dissensus

SUMMARY:
Deep brain stimulation (DBS) has become a cornerstone therapy for advanced Parkinson's disease (PD), showing superior outcomes over best medical treatment in randomized clinical trials. By delivering adjustable electrical stimulation to key basal ganglia targets, DBS improves tremor, rigidity, bradykinesia, and motor fluctuations, while also reducing dopaminergic medication requirements. Its success, however, depends not only on precise surgical targeting but also on careful patient selection, multidisciplinary planning, and structured long-term follow-up.

In Italy, PD affects nearly 176,000 individuals, of whom an estimated 2-4.5% are potential candidates for DBS. A national survey conducted by the Italian Neurosurgery Society (SINch) revealed marked heterogeneity in surgical approaches, target selection, and team composition across DBS centers-reflecting similar international variability. Yet, clear national indications and guidelines have not been established. To address this gap, we conducted an expert consensus using the Delphi methodology.

DETAILED DESCRIPTION:
Deep brain stimulation (DBS) has become a cornerstone therapy for advanced Parkinson's disease (PD), consistently showing superior outcomes over best medical treatment in randomized clinical trials. By delivering adjustable electrical stimulation to specific basal ganglia targets, DBS provides sustained improvement in cardinal motor symptoms such as tremor, rigidity, and bradykinesia, while also mitigating motor fluctuations and dyskinesias. It often enables a substantial reduction in dopaminergic medication requirements, thereby decreasing treatment-related side effects and improving quality of life. Nonetheless, the success of DBS relies not only on accurate surgical targeting but also on careful patient selection, multidisciplinary planning, and long-term follow-up.

In Italy, PD affects nearly 176,000 individuals, of whom an estimated 2-4.5% may be suitable candidates for DBS. Despite this, effective implementation remains challenging. A national survey by the Italian Neurosurgery Society (SINch) revealed marked heterogeneity among DBS centers, particularly in surgical approaches, target selection, perioperative protocols, and team composition. While such variability mirrors international patterns, in Italy it is compounded by the absence of nationally endorsed guidelines or standardized care pathways. This lack of uniformity risks inequities in access, indications, and outcomes, raising concerns about quality of care and resource allocation within the national healthcare system.

Developing clear, evidence-based recommendations is therefore of paramount importance. Standardized indications and procedural frameworks would support patient selection, harmonize surgical practice, and guide multidisciplinary teams in delivering high-quality long-term care. Moreover, national guidelines would facilitate benchmarking across centers, promote training and education, and ensure equitable access to state-of-the-art treatment for all eligible patients.

To address these needs, we convened a panel of Italian experts in functional neurosurgery. Using the Delphi consensus methodology, we systematically gathered, refined, and integrated expert opinions on key aspects of DBS therapy for PD, with the aim of establishing practical, consensus-based recommendations tailored to the Italian healthcare setting.

ELIGIBILITY:
Panelist selection

Healthcare professionals will be recruited as panelists based on the following predefined criteria:

Inclusion criteria:

* At least 5 years of clinical experience in the care of patients with Parkinson's disease, including involvement in deep brain stimulation (DBS) implantation (in both teaching and non-teaching settings).
* Prior participation in guideline development or authorship of at least one peer-reviewed publication on neuromodulation in Parkinson's disease.

Exclusion criteria:

- None.

Recruitment strategy:

- Purposive sampling will be applied to identify Italian panelists, primarily through a review of recent publications in the field of DBS for Parkinson's disease. Panelist selection will adhere to the predefined criteria, with deliberate efforts to ensure gender balance and broad geographical representation across Italy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare professionals representing italian neurosurgeons with expertise in the field of deep brain stimulation of patients with Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Consensus use of Deep Brain Stimulation in Parkinson's Disease | 3-6 months
  A diverse panel of experts from across Italy, identified through pre-specified qualification criteria, will participate in iterative Delphi rounds to develop consensus on the indications and parameters of deep brain stimulation for Parkinson's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Anesthesia and Intensive Care, Magna Graecia University, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No
Due to the study design (expert consensus), individual patient data do not require to be shared